CLINICAL TRIAL: NCT05614570
Title: SSVEP Evaluation of Brain Function
Status: Completed | Type: Observational
Sponsor: Headsafe MFG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-10-891
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic brain injury; Concussion; Steady state visual evoked potential; Electroencephalography; Sports Concussion; Sports Medicine
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Baseline: This cohort contains individuals tested at baseline, usually in the pre-season of their sporting season
  Interventions: Device: SSVEP Device; Other: SCAT5
- Concussed: This cohort contains individuals who have had a concussion, diagnosed by a doctor.
  Interventions: Device: SSVEP Device; Other: SCAT5

INTERVENTIONS:
Device: SSVEP Device — Non-invasive, non-interventional SSVEP sensor device
  Other Names: Nurochek
Other: SCAT5 — The Sport Concussion Assessment Tool version 5

SUMMARY:
The investigational device used in this clinical investigation, the Nurochek Headset, is a portable electroencephalogram (EEG) headset which delivers a visual stimulus and measures a VEP. The visual stimulus is delivered to the subjects' eyes via light-emitting diodes, and the EEG measures the user's visual-evoked potential. This headset communicates with an application on a smartphone which processes the signals and transmits them to a secure cloud server for analysis and storage of the data.

The primary objective of this clinical investigation was to evaluate the performance of the investigation device (NCII) against clinical diagnosis and SCAT 5, in the accurate detection of mild traumatic brain injury (mTBI). The primary endpoint outlined for this study was set at the collection of 100 valid investigational device readings from individuals with concussion

The aim of this study was to collect data from 100 readings from individuals with concussion. It was estimate that approximately 10-20% of baselined players would suffer a concussion during the season. There it was estimated there would be a need to baseline 500-1000 individuals in order to achieve the number of concussions required. The initial assumption was that sites would provide players pre-season and make players available for testing post-concussion. In practice, some sites provided player data only post-concussion event (such as medical clinics). Participants were required from sporting clubs, medical clinicals and schools.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 14 years and older, participating in sport-related activities.

Exclusion Criteria:

* Individuals were excluded if they had a history of seizures, history of epilepsy, structural brain injuries, legal blindness, or sensitivity to flashing lights.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population contained individuals 14 years or older who play sport. They were requited from a large variety of sport types and facilities including local clubs, medical centres and schools.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Steady State Visual Evoked Potential | 30 days
  A measure of the steady state visual evoked potential (SSVEP) from the device
SCAT5 Score | 30 days
  The score from the SCAT5 as determined at Step 6.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Donaldson, MBBS, Principal Investigator — Principal Investigator
Locations (1):
- Headsafe, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No